CLINICAL TRIAL: NCT05411068
Title: Reliability And Validity Of Urdu Version Of Disabilities Of The Arm, Shoulder And Hand Questionnaire Among Carpal Tunnel Syndrome Patients
Brief Title: Reliability And Validity Of Urdu Version Of Disabilities Of The Arm, Shoulder And Hand Questionnaire
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00271
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Disabilities Of The Arm, Shoulder And Hand Questionnaire; Urdu Version; Reliability; Validity; Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of study is to convert Disabilities Of The Arm, Shoulder And Hand Questionnaire into Urdu and test its reliability and validity among the Pakistani citizens. Also check its correlation with Boston carpal tunnel syndrome questionnaire and visual analogue scale as well.

DETAILED DESCRIPTION:
A cross-sectional study will be conducted after approval from ethical review committee of Riphah international university of Faisalabad. Total of 90 participants will be included in this study from different community areas, hospitals and rehabilitation centers with carpal tunnel syndrome. 71 of them will be male and 19 will be female. Disabilities of the Arm, Shoulder, and Hand questionnaire will be correlated with Boston carpal tunnel syndrome questionnaire and visual analogue scales. These questionnaires will be filled by participants firstly for baseline, secondly after treatment and third one week later as a follow up. Written informed consents will be taken before filling questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Subjects with phalen's and Tinnel's test positive.

Exclusion Criteria:

Participants who had following conditions:

* Diabetes mellitus, thyroid disease, rheumatoid arthritis, radiculopathy of cervical spine, cognitive impairment.
* Hand surgery within previous 3 months.
* Difficulty in understanding of language.
* Musculoskeletal disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Carpal tunnel syndrome population of Pakistan will be included in study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Disabilities Of The Arm, Shoulder And Hand Questionnaire | 1st day
  Disabilities Of The Arm, Shoulder And Hand Questionnaire scale was designed to identify musculoskeletal disorders in the upper limbs, however it is also an appropriate outcome measure for Carpal Tunnel Syndrome. Disabilities Of The Arm, Shoulder And Hand Questionnaire questionnaire has 30 questions. These questions assess how difficult it is to execute a variety of functions due to arm, shoulder, or hand issues (21 items). They also look at intensity of symptoms (5 items), as well as psychological impact of condition (4 items).There are five response possibilities for each item, varying from little difficulty or no symptoms (1 point) to unable to do activity or severe condition (5 points).
Boston carpal tunnel syndrome questionnaire | 1st day
  Boston carpal tunnel syndrome questionnaire is divided into two sub-scales: symptom severity & functional status. Every question has a 5-point scale, with 1 indicating no difficulties and 5 indicating significant symptoms or reduced function. Boston carpal tunnel syndrome questionnaire is a brief questionnaire that may be completed in 10 minutes.
Visual analogue scale | 1st day
  Visual analogue scale is a tool which is used to measure pain severity. It ranges from 0-10 with 0 means no pain ranges between 1 to 3 mean mild pain, 4 to 6 represents moderate pain and 7 to 9 means severe pain whereas 10 means unbearable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No